CLINICAL TRIAL: NCT05657769
Title: A Randomized Trial of Preventive Care System Application Effectiveness on the Treatment of Diabetic Patients in Bandung
Brief Title: Preventive Care System Application Effectiveness Study on the Treatment of Diabetic Patients in Bandung
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PT Bio Farma (Industry)
Collaborators: Immanuel Hospital (Unknown); Prodia the CRO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Medwell-01-2022
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study is conducted with the primary hypothesis that the diabetes treatment with Medwell intervention can significantly reduce the HbA1c level better than without Medwell intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Treatment) (Experimental): Regular diabetes treatment with additional Medwell application and wearable device.
  Interventions: Device: Medwell Preventive Care Application
- Group II (Control) (Active Comparator): Regular diabetes treatment only with a diary card to record daily activities manually.
  Interventions: Device: Manual Records

INTERVENTIONS:
Device: Medwell Preventive Care Application — Regular diabetes treatment with additional Medwell application and wearable device.
  Arms: Group I (Treatment)
Device: Manual Records — Regular diabetes treatment only with a diary card to record daily activities manually.
  Arms: Group II (Control)

SUMMARY:
Randomized, unblinded, controlled, two arms parallel group, prospective intervention study

DETAILED DESCRIPTION:
The objective of the study is to compare the progression of HbA1c in diabetic patients after applying a Medwell digital application in addition to regular diabetes treatment (treatment arm) with regular diabetes treatment of diabetic subjects alone (control arm).

The primary endpoint will be measured as the difference between 3 months HbA1c relative to baseline in eligible subjects. Normally, HbA1c in each subject is expected to either stable or slightly increase overtime. In this study we are interested in measuring the difference in HbA1c 3 months post randomization. It is expected that in the experimental arm, HbA1c will slightly decrease, while in the standard arm, HbA1c will either remain the same or will slightly increase after 3 months in the study. Previous study shows that the standard deviation of the difference in HbA1c within 1 year is 0.97%.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are in the diabetes type 2 status (based on Perkeni standard) HbA1c is ≥6.5%
* Aged 18 - 60 years old
* Have compatible smartphone (minimum android 8 or iOS 13) and internet connection
* Receiving regular diabetes treatment
* Giving consent and commitment to participate in the study until finish
* Located in Bandung Area within the treatment period (up to 3 month after receiving the treatment)
* Subject is determined to be able to complete daily physical activities.

Exclusion Criteria:

* Pregnant (based on test pack)
* Participation in other weight loss program
* Use of other tracking application
* Having any abnormalities that affecting blood erythrocyte age defined by laboratory examination
* Have other severe diabetic complications that prevent subjects from participating in the prescribed program (Such as stroke, cardiac diseases (CHF stage III-IV), COPD or asthma with acute exacerbation and other respiratory diseases, peripheral artery disease, CKD stage 3-5) and other severe diseases that by the investigator's judgment, could not participate in this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-11-12 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
HbA1C Changes | 3 months
  Change in HbA1c from baseline to month 3 for all groups.
  Change in HbA1c from baseline to month 3 for all groups.
  Change in HbA1C from baseline to moth 3 of all group

SECONDARY OUTCOMES:
Evaluate the exercise | 3 months
  Mean weekly frequency of exercise
Evaluate the exercise | 3 months
  Proportion of exercise prescribed by physicians timely performed by subjects
Evaluate the exercise | 3 months
  Mean duration of each exercise
Drug Adherence | 3 months
  Proportion of administered drugs timely consumed by subjects
Anthropometry I (BMI) | 3 months
  Change in the BMI after 3 months
Anthropometry II (Body Fat) | 3 months
  Change in the Body Fat after 3 months
Anthropometry III (Muscle Mass) | 3 months
  Change in the Muscle Mass after 3 months
Lab outcome I (Fasting glucose) | 3 months
  Change in the lab measurement from baseline to month 3 for fasting glucose
Lab outcome II (2 hours post prandial glucose) | 3 months
  Change in the lab measurement from baseline to month 3 for 2 hours postprandial glucose
Lab outcome III (total cholesterol) | 3 months
  Change in the lab measurement from baseline to month 3 for total cholesterol
Lab outcome IV (low density lipoprotein) | 3 months
  Change in the lab measurement from baseline to month 3 for low density lipoprotein
Lab outcome V (high density lipoprotein) | 3 months
  Change in the lab measurement from baseline to month 3 for high density lipoprotein
Lab outcome VI (triglyceride) | 3 months
  Change in the lab measurement from baseline to month 3 for triglyceride

CONTACTS AND LOCATIONS:
Overall Officials: Ratih Nursiana, Principal Investigator — RS Immanuel; Indahwaty Indahwaty, Study Director — RS Immanuel
Locations (1):
- Immanuel Hospital, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No